CLINICAL TRIAL: NCT03678480
Title: A Phase 2, Randomized, Double-Blind Study of HTD1801 vs Ursodeoxycholic Acid (UDCA) in Adolescents With Primary Sclerosing Cholangitis (PSC)
Brief Title: A Study of HTD1801 in Adolescents With Primary Sclerosing Cholangitis (PSC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Corporate decision
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTD1801.PCT006
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2020-07

CONDITIONS: Primary Sclerosing Cholangitis; Cholangitis; Cholangitis, Sclerosing; Bile Duct Diseases; Biliary Tract Diseases; Digestive System Diseases; Adolescent
MeSH Terms: conditions — Cholangitis, Sclerosing; Cholangitis; Bile Duct Diseases; Biliary Tract Diseases; Digestive System Diseases | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HTD1801 500 mg BID (twice daily), or 1000 mg/day (Experimental): HTD1801 tablets in double-blind capsules, 250 mg
  Interventions: Drug: HTD1801
- Ursodeoxycholic Acid (UDCA) 250 mg BID, or 500 mg/day (Active Comparator): UDCA tablets in double-blind capsules, 250 mg
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: HTD1801 — HTD1801 capsules, 250mg
  Arms: HTD1801 500 mg BID (twice daily), or 1000 mg/day
Drug: Ursodeoxycholic Acid — UDCA capsules, 125mg
  Arms: Ursodeoxycholic Acid (UDCA) 250 mg BID, or 500 mg/day

SUMMARY:
Randomized, double-blind, active-controlled, parallel-group study of HTD1801 in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 35 kg
* Previous cholangiographic evidence of PSC by magnetic resonance cholangiopancreatography (MRCP) or direct cholangiography or liver biopsy findings
* Serum GGT ≥ 2 × upper limit of normal (ULN)
* On a stable UDCA treatment regimen for ≥ 8 weeks

Exclusion Criteria:

* Secondary sclerosing cholangitis
* Percutaneous or endoscopically-placed biliary drain or stent
* History of cholangiocarcinoma or clinical suspicion of new dominant stricture within 1 year
* Ascending cholangitis requiring intravenous antibiotic therapy within 60 days prior to Screening
* Concomitant overlap syndrome with primary biliary cholangitis (PBC)
* Significant hepatic decompensation
* Alternative causes of chronic liver disease
* Hospitalization for colitis within 30 days prior to Screening
* Serum creatinine > 1.2 x ULN
* Hemoglobin < 10 g/dL
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-10-04 (Estimated); Study Completion 2021-11-04 (Estimated)

PRIMARY OUTCOMES:
change in gamma-glutamyl transferase (GGT) | 18 weeks

SECONDARY OUTCOMES:
percentage of patients whose GGT normalizes to <50 units/liter | 18 weeks
change in aspartate aminotransferase (AST) | 18 weeks
change in alanine aminotransferase (ALT) | 18 weeks
change in alkaline phosphatase (ALP) | 18 weeks
change in total bilirubin | 18 weeks
change in C-reactive protein (CRP) | 18 weeks
incidence of adverse events | 18 weeks

IPD SHARING:
Plan to Share IPD: No